CLINICAL TRIAL: NCT03173612
Title: The Efficiency of CAMS-2016 Trial for the Newly Diagnosed Pediatric Acute Myeloid Leukemia: A Prospective Single Centre Trial From China
Brief Title: The Efficiency of CAMS (Chinese Academy of Medical Sciences)-2016 Trial for Pediatric Acute Myeloid Leukemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Zhu Xiaofan, Director, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML-CAMS-2016
Record Dates: First submitted 2017-05-16; First posted 2017-06-02 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Dasatinib; Idarubicin; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AML-CAMS-2016 trial (Experimental): AML-CAMS-2016 regimen includes risk-stratified therapy and the use of Dasatinib in CBF-AML.The induction regimen includes MAE (etoposide 150mg/㎡/d d1-5, cytarabine 200mg/㎡/d d6-12 , mitoxantrone 5 mg/㎡/d d6-10), CAG (aclacinomycin 6mg/㎡/d d1-8, Ara-C 10mg/㎡ q12h d1-14 , G-CSF 200ug/㎡/d d1-14),IAE (idarubicin 8 mg/㎡/d d1-3, Ara-C 500mg/㎡/d d1-3 d8-10, VP-16 200mg/㎡/d d8-10).Consolidation regimen includes IA (Ara-C 1g/㎡ q12h d1-4, IDA 10mg/㎡/d d1), MA (Ara-C 1g/㎡ q12h d1-4, MTZ 5mg/㎡/d d1-3), IAE (IDA 10mg/㎡/d d1, Ara-C 3g/㎡ q12h d1-3, VP-16 100mg/㎡/d d1-5), MAE (Ara-C 200mg/㎡ d4-8, VP-16 150mg/㎡/d d1-3, MTZ 5mg/㎡/d d4-6),EA (Ara-C 2g/㎡ q12h d1-5, VP-16 100mg/㎡/d d1-5),IAE (IDA 10mg/㎡/d d1, Ara-C 3g/㎡ q12h d1-3, VP-16 100mg/㎡/d d1-5),EA (Ara-C 2g/㎡ q12h d1-5, VP-16 100mg/㎡/d d1-5),MAE (Ara-C 200mg/㎡ d4-8, VP-16 150mg/㎡/d d1-3, MTZ 5mg/㎡/d d4-6). Dasatinib (60-80mg/㎡) is used in CBF-AML as a part of consolidation therapy.
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Primary AML includes CBF-AML and non-CBF-AML. Children with a WBC (white blood cell) lower than 4,000/μL and low proliferative bone marrow at diagnosis are treated with CAG. Other children are treated with MAE. The rescue regimen for children who showed M3 marrow after MAE or CAG is IAE. Consolidation therapy consisted of four (for CBF-AML) or five (for non-CBF-AML) courses, and triplein trathecal therapy is given as a part of each course. After the second course of therapy, CBF-AML are stratified into two risk groups, while non-CBF-AML patients in remission are stratified into three risk groups.Consolidation regimen for CBF-AML includes IA, MA, IA, MA. Dasatinib is used in CBF-AML as a part of consolidation therapy. Consolidation regimen for non-CBF-AML includes IAE, MAE, EA, IAE, EA or MAE.
  Other Names: cytarabine(Ara-C); etoposide(VP-16); idarubicin(IDA); aclacinomycin(Acla); granulocyte colony-stimulating factor(G-CSF); Mitoxantrone

SUMMARY:
The purpose of this study is to evaluate that whether the AML (acute myeloid leukemia)-CAMS (Chinese Academy of Medical Sciences)-2016 regimen, includes risk-stratified therapy and the use of Dasatinib in CBF (Core binding factor)-AML, can improve the outcome in childhood AML.

DETAILED DESCRIPTION:
Primary AML includes CBF(Core binding factor)-AML and non-CBF-AML. After the second course of therapy, CBF-AML are stratified into two risk groups: low-risk children are defined as those with CR after MAE or CAG, high-risk children are those with CR after consolidation course 1 or IAE. Non-CBF-AML patients in remission are stratified into three risk groups: low-risk children are defined as those with t(1；11)(q21；q23) , GATA1, NPM1/IDH1/IDH2 without FLT3/ITD,or an age younger than 2 years without high-risk factors; high-risk children are those with CR after consolidation course 1 or IAE or with abnormalities of monosomy 7, 5q- , t(16;21), t(9;22) (Philadelphia chromosome [Ph1]), FLT3/ITD,-17/TP53, RPN1-MECOM, RUNX1-EVI1, MLF1-NPM1, PRDM16-RPN1, DEK-NUP214, ETV6(TEL)-HLXB9(MNX1), NUP98-NSD1; intermediate-risk children are those who were not in either a low-risk or high-risk group.Low-risk children were treated only with chemotherapy, regardless the availability of a suitable HSCT donor. All high-risk children were allocated to Allo-hematopoietic stem cell transplantation (HSCT) in the first remission, including unrelated bone marrow transplantation (BMT). Auto-HSCT is recommended for intermediate-risk children. No prophylactic cranial irradiation is included in the protocol. Patients are treated on an inpatient basis during each treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosis of de novo Acute Myeloid Leukemia

Exclusion Criteria:

* Children with Down's syndrome and acute promyelocytic leukemia, hybrid acute leukemia

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Estimated)
Dates: Start 2016-08; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Complete remission | through study completion, an average of 7 year
  Fewer than 5% blast cells in the bone marrow aspirate and the absence of extramedullary involvement (EMI)
Overall Survival (OS) | From date of diagnosed until the date of death from any cause, assessed up to 60 months
  Overall Survival
Event-free Survival (EFS) | From date of diagnosed until the date of first relapse or date of death from any cause, whichever came first, assessed up to 60 months
  Event-free Survival
Disease-free Survival (DFS) | From date of remission until the date of first relapse or date of death from any cause, whichever came first, assessed up to 60 months
  Disease-free Survival

SECONDARY OUTCOMES:
all cause mortality | one year after diagnosed
  Dead during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Xiaofan, Study Chair — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- InstituteHBDH, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided